CLINICAL TRIAL: NCT03820037
Title: A Phase I, Open-Label, Randomised, Three-Period, Three-Sequence, Partial Replicate Crossover Study to Investigate the Relative Bioavailability and Bioequivalence of Opicapone Obtained From Two Different Sources, Under Fasting Conditions After Single-dose Administration in Healthy Subjects
Brief Title: Relative Bioavailability and Bioequivalence of Opicapone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-132
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPC, Ongentys (Active Comparator): Single oral doses of 50 mg opicapone, administered using the reference (Ongentys ®) active pharmaceutical ingredient (API) source
  Interventions: Drug: Ongentys
- BIA 9-1067 (Experimental): Single oral doses of 50 mg opicapone, administered using the test (BIA 9-1067)
  Interventions: Drug: BIA 9-1067 (test)

INTERVENTIONS:
Drug: Ongentys — single oral 50 mg (capsule containing 50 mg OPC) under fasting conditions
  Arms: OPC, Ongentys
Drug: BIA 9-1067 (test) — single oral 50 mg (capsule containing 50 mg OPC) under fasting conditions
  Arms: BIA 9-1067

SUMMARY:
the purpose assess the relative bioavailability and bioequivalence of two active pharmaceutical ingredient (API) sources of opicapone (OPC, Ongentys® and BIA 9-1067) following single 50 mg dose administration under fasting conditions in healthy volunteers

DETAILED DESCRIPTION:
This will be a Phase I, open label, randomized, partial-replicate, three-period, three-sequence crossover study to investigate the relative bioavailability and bioequivalence of 2 API sources of OPC (BIA 9-1067 [Test] and Ongentys® [Reference]) in healthy adult subjects.

Subjects will be randomized in a 3-period, 3-sequence crossover design; each subject will receive 2 single oral 50 mg doses of the Reference API source of OPC, and a single 50 mg dose of the Test API source of OPC under fasting conditions.

Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the first dose administration. Subjects will be admitted into the Clinical Research Unit (CRU) on Day 1 and be confined to the CRU until discharge on Day 3. There will be a washout period of at least 14 days between each dose. A follow-up visit will be performed 7 to 14 days after dosing in the last treatment period or early discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, between 18 and 55 years of age, inclusive.
2. Body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive.
3. Healthy subjects as determined by no clinically significant findings from medical history, physical examination, complete neurological examination, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhaemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at Screening and Check in as assessed by the Investigator (or designee).
4. Females will not be pregnant (i.e. the the pregnancy test at screening and at admission to each treatment period must be negative), or lactating, and females of childbearing potential and males will agree to use contraception.
5. Able to comprehend and willing to sign and date an Informed Consent Form (ICF) before any study-specific screening procedure is performed, and to abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, lymphatic, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, genitourinary, immunological, connective tissue diseases or disorders, musculoskeletal, psychiatric disorder, or have a clinically relevant surgical history as determined by the Investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
3. History of febrile illness within 10 days prior to the each dose of study drug, or subjects with evidence of active infection
4. Acute gastrointestinal symptoms (eg nausea, vomiting, diarrhoea, heartburn) as determined by the Investigator (or designee).
5. Significantly impaired hepatic function, defined as any of the following (confirmed by repeat):

   1. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 x upper limit of normal (ULN)
   2. Total bilirubin (TBL) > 2 x ULN
6. Significant personal or family history of haemostatic disorders
7. History of galactose intolerance (eg the Lapp lactase deficiency or glucose-galactose malabsorption)
8. Symptomatic orthostatic hypotension (drop of > 20 mmHg in systolic blood pressure and/or > 10 mmHg in diastolic blood pressure) when moving from supine to standing position, together with other symptoms, e.g., dizziness.
9. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
10. History of alcoholism or drug/chemical abuse within 2 years prior to Check in to the first treatment period.
11. Alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
12. Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at Screening or Check in to each treatment period.
13. Positive hepatitis panel and/or positive human immunodeficiency virus test
14. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to first dose of study drug.
15. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to Check-in of the first treatment period, unless deemed acceptable by the Investigator (or designee).
16. Use or intend to use any prescription medications/products within 14 days prior to dosing, unless deemed acceptable by the Investigator (or designee).
17. Use or intend to use slow release medications/products considered to still be active within 14 days prior to Check in, unless deemed acceptable by the Investigator (or designee).
18. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 7 days prior to Check in, unless deemed acceptable by the Investigator (or designee).
19. Use of tobacco or nicotine containing products within 3 months prior to Check in, or positive cotinine at Screening or Check-in.
20. Receipt of blood products within 2 months prior to Check in.
21. Donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
22. Subjects who are vegetarians, vegans or have medical dietary restrictions
23. Poor peripheral venous access.
24. Have previously completed or withdrawn from this study or any other study investigating opicapone, and have previously received the investigational product.
25. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-06-09 (Actual); Study Completion 2019-06-09 (Actual)

PRIMARY OUTCOMES:
area under the plasma concentration-time curve from time zero to infinity (AUC0 ∞) | Day 1 up to day 14
  PK parameters from Blood samples to be be collected for the analysis of plasma concentrations of opicapone.
area under the plasma concentration-time curve from time zero to the last observable concentration at time t (AUC0 t) | Day 1 up to day 14
  PK parameters from Blood samples to be be collected for the analysis of plasma concentrations of opicapone.
maximum observed plasma concentration (Cmax) | Day 1 up to day 14
  PK parameters from Blood samples to be be collected for the analysis of plasma concentrations of opicapone.

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided